CLINICAL TRIAL: NCT05453175
Title: The Effect of Uninterrupted and Interrupted Sitting on Vascular Health and Cognitive Function in People with Long COVID-19
Brief Title: Uninterrupted and Interrupted Sitting in Long COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Winchester (Other)
Collaborators: University of Gloucestershire (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: UoW_Faulkner_LCOVID_22
Record Dates: First submitted 2022-07-11; First posted 2022-07-12 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interrupting sitting (Experimental): Participants will engage in low intensity physical activity every thirty minutes up to 120 minutes
  Interventions: Other: Interrupting sitting with Physical activity
- Control (No Intervention): Participants will remain seated for the entire 120 minutes

INTERVENTIONS:
Other: Interrupting sitting with Physical activity — Participants will engage in three minutes of walking, five sit to stands and five calf raises every thirty minutes
  Arms: Interrupting sitting

SUMMARY:
People who sit uninterrupted for prolonged periods time have been shown to have poorer cardiovascular health compared to those that regularly interrupt it (e.g. standing up and moving). Cognition and brain function has also been shown to be impaired following uninterrupted sitting. Research has shown that interrupting sitting with exercise improves cardiovascular health in healthy men and women cognition, feeling of fatigue and cerebral oxygenation. Low intensity physical activity can help people with Long coronavirus disease (COVID) by reducing feelings of fatigue.

Individuals with long COVID have symptoms such as fatigue and brain fog. As such, people with long COVID may spend more time sitting during the day and demonstrate worsened cardiovascular and cognitive health. As such, there may be greater levels of cognitive decline and worsened cardiovascular health outcomes. In this study the investigators are interested in assessing the cardiovascular health and brain function of people with (and without) long COVID before and after uninterrupted and interrupted sitting.

Interruptions will be every 30 minutes during a 120 minute sitting period. Interruptions are self-paced and include up to three minutes of walking, five heel raises and five sit-to-stands at each interruption. To ensure external validity of the project, all interruptions are functional activities which can be reproducible in a home environment. Vascular health and cognitive function will be assessed before and after the interrupted and uninterrupted trials. Eligible participants will be aged over 18 years, have displayed symptoms of long COVID for more than 4 weeks, and have been diagnosed with long COVID via their GP or through a long COVID clinic. Involvement in the study will include three visits to a physiology laboratory at the University of Winchester or University of Gloucestershire. Involvement can be expected to last up to 40 days to account for the necessary time required between laboratory visits.

DETAILED DESCRIPTION:
Design:

The present study will be a laboratory study. The intervention group being persons suffering from Long COVID, and the control group being a healthy aged match group. Both the experimental and control groups will be randomised into either performing uninterrupted or interrupted sitting first to reduce the risk of order and learning effects associated with the trials. All individuals who are identified from general practitioner (GP) practices (e.g. Park and St Francis Surgery, Chandlers Ford near Winchester or associated surgeries and clinics) or long COVID clinics (e.g. Gloucestershire Health and Care NHS (National Health Service) Foundation Trust, Post Covid Syndrome Service and Southampton and Isle of Wight Long Covid Clinic, Solent NHS Trust, Southern Health NHS Trust and Isle of Wight NHS Trust), who meet the inclusion criteria will be provided with equal opportunity to engage with the study provided they are able to travel to either the University of Winchester or University of Gloucestershire for assessment. Healthy participants who will form the control group will also have equal opportunity to engage with the study providing they meet the inclusion criteria and are able to travel to either the University of Winchester or University of Gloucestershire for assessment.

The purpose and design of this study has been discussed with all members of the study team, and at a Patient and Public Involvement (PPI) meeting, with people currently suffering from Long COVID.

Recruitment:

Potential participants will initially be identified by the healthcare team at Park and St Francis Surgery, the Gloucestershire Health and Care NHS Foundation Trust, Post Covid Syndrome Service, Southampton and Isle of Wight Long Covid Clinic, Solent NHS Trust, Southern Health NHS Trust and Isle of Wight NHS Trust or associated surgeries and clinics according to study inclusion/exclusion criteria. The clinical team will gain documented verbal consent from potential participants for their contact details to be provided to the research team at the University of Winchester (Prof. James Faulkner, Dr Helen Ryan-Stewart and Mr Nick Hudson) and University of Gloucestershire (Dr Simon Fryer, Dr Keeron Stone and Mr Callum Thomas) who will then contact patients directly to discuss their potential participation.

As described above (Design), the research team will make every effort to provide all participants a fair and equal opportunity to engage with the study provided they are able to travel to the University sites for study participation.

Informed Consent:

Participants will be provided with a study information sheet which outlines their possible involvement and will have opportunities to discuss the study with the research team prior to deciding as to whether to participate or not. Each participant will have had sufficient time (>24-hours) to read the information sheet and will be able to ask questions to the research team both by phone prior to attending their first assessment visit and upon arrival to the Exercise Physiology Laboratory at the University of Winchester or University of Gloucestershire before providing voluntary written consent for participation in this study. Participants will be reminded that they can withdraw from the study at any time and without repercussion of any kind.

Procedures:

All participants will complete an adapted health history questionnaire and the EQ-5D-5L quality of life questionnaire during familiarisation. Participants will be fitted with an activity monitor for seven days following familiarisation to attain measures of physical activity/sedentary behaviour during a typical week. Participants with long COVID will be asked to complete a series of questionnaires which measure the type and severity of their symptoms as well as their functional status (COVID-19 Yorkshire Rehabilitation tool, COVID-19 symptom score, Post COVID-19 Functional Status Scale). Central and peripheral blood pressure, pulse wave velocity, cognitive function and cerebral perfusion will be measured in a supine and seated position at baseline and following 120 minutes of interrupted or uninterrupted sitting. Central and peripheral blood pressure, pulse wave velocity and cerebral perfusion will be measured while seated during the sitting period. Following visiting the laboratory, long COVID participants will complete the DePaul Symptom Questionnaire Post-Exertional Malaise (DSQ-PEM) and receive a telephone call from the research team within 72 hours of their visit. Should participants present symptoms of PEM, their participation in future visits to the laboratory will be delayed. Should symptoms of PEM persist for 30 days they will be withdrawn from the study and their GP will be contacted.

Confidentiality:

Participants will be assured of the confidentiality of the research process. All data will be anonymised using alpha- numeric code which will be stored on a password protected network, accessible by only the named researchers involved with the study. Hard copies of data will be locked in a filing cabinet in the office of Prof. James Faulkner in Centre for Sport of the University of Winchester's King Alfred campus and in Dr Simon Fryer's locked office at the Oxstalls campus at the University of Gloucestershire. Physical copies of data will not be removed from these offices. Due to collaboration, data will need to be shared between institutions. Data will be uploaded to a secure, password protected folder on Microsoft OneDrive. All data will be presented as group means and standard deviations. All data will be kept for 7 years, with Prof. Faulkner and Dr Fryer responsible for its security during this time and its appropriate disposal once this period has elapsed.

Risks/Burdens:

Potential risks to participants could be caused by over exertion during a physical activity intervention within the experimental condition. To minimise this risk, the type and intensity of physical activity chosen is low and comfortable to complete for participants with low levels of mobility and who experience fatigue after minimal activity. Participants will have up to 30 days between visits to further minimise any risks. In addition, participants will undertake the Covid 19 Yorkshire Rehab Screen (C19-YRS). This will allow the researchers to gain prior knowledge of participants level of fatigue, mobility, and cognitive function prior to involvement in the study and participant selection.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COVID-19 (via the NHS by polymerase chain reaction (PCR)/lateral flow positive results or by clinical diagnosis based on set criteria)
* Clinical diagnosis of Long COVID, reported by a GP, defined as 'signs and symptoms that develop during or following an infection consistent with COVID-19 which continue for more than 4 weeks and are not explained by an alternative diagnosis' (NICE guidelines, October 2020).
* Minimum age of 18 years
* Cognitively aware of task demands

Exclusion Criteria:

* Unable to undertake necessary physical activity for the study Unable to remain seated for 120 minutes at a time Unstable cardiovascular conditions
* People with diabetes
* People with dementia
* Recent (previous 6 months) moderate to severe injury of the lower extremities
* No positive COVID test or signs and symptoms within 6 weeks for healthy control
* No positive COVID test within 4 weeks for Long COVID group

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Pulse Wave Velocity | Change from baseline to 120 minutes post baseline
  Carotid femoral pulse wave velocity (PWV) using SphygmoCor XCEL. Lower numbers represent healthier PWV, and in turn better vascular health

SECONDARY OUTCOMES:
Central and peripheral pulse wave analysis | Change from baseline to 120 minutes post baseline
  A non-invasive method of measuring blood pressure, arterial stiffness, how much time the heart spends pumping, and the ability of the arterial system to meet the heart's energy requirements
Cognitive function | Change from baseline to 120 minutes post baseline
  A two part cognitive assessment completed on an IPad using visual screening and working memory. Scores that are lower in time (seconds) and errors indicate better performance at the task
Quality of Life - EuroQuol 5 Dimensions 5 levels (EQ-5D-5L) | Baseline
  5-item questionnaire that assesses quality of life. Higher scores mean better quality of life. Minimum score is 1 and the maximum score is 5 for each dimension

OTHER OUTCOMES:
DePaul Symptom Questionnaire: Post-Exertional Malaise (DSQ-PEM) | Up to 72 hours, and weekly (up to 4 weeks) following each laboratory visit
  The DSQ-PEM is a 10 item questionnaire used to assess presence of post-exertional malaise based on the frequency and severity of symptoms. Items are scored from 0 to 4, with 0 relating to a low value and 4 relating to a high value.

CONTACTS AND LOCATIONS:
Overall Officials: James Faulkner, PhD, Principal Investigator — University of Winchester
Locations (1):
- Park and St Francis, Winchester, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individuals wanting access to IPD should contact the lead investigator (James.Faulkner@winchester.ac.uk).
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Starting after 6 months of publication
Access Criteria: Available to all researchers interested in long covid research